CLINICAL TRIAL: NCT01177826
Title: Case-control Study to Evaluate the Vaccine Effectiveness of GlaxoSmithKline (GSK) Biologicals' Live Attenuated Human Rotavirus (HRV) Vaccine (Rotarix™) Against Community-acquired Rotavirus Severe Gastroenteritis (RV SGE) Among Hospitalised Children Born After 1 October 2006, in Belgium
Brief Title: Effectiveness Study of GSK Biologicals' Rotarix TM Vaccine in Hospitalized Children
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111426
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Infections, Rotavirus; Rotavirus Vaccines
Keywords: Hospitalized; Rotavirus; Children; effectiveness; Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples

GROUPS / COHORTS (2):
- Group 1: Cases
  Interventions: Procedure: Sample collection
- Group 2: Controls
  Interventions: Procedure: Sample collection

INTERVENTIONS:
Procedure: Sample collection — Stool sample

SUMMARY:
The purpose of this study is to assess vaccine effectiveness of Rotarix in preventing rotavirus severe gastroenteritis among hospitalized infants, in Belgium.

ELIGIBILITY:
Inclusion Criteria:

For confirmed cases:

* A male or female child born after 01 October 2006 and at least 14 weeks of age at the time of hospital admission.
* Child admitted at the study hospital for SGE during the study period.
* Onset of SGE ≤ 14 days prior to admission.
* Written informed consent obtained and signed from the parent or guardian of the child.
* Stool samples collected during the first 48 hours of hospitalisation and then tested positive for RV by PCR.

For controls:

* A male or female child born after 01 October 2006 and at least 14 weeks of age at the time of the hospital admission or visit to the hospital outpatient clinic.
* Hospitalised or visiting the hospital outpatient clinic for non-GE causes at the same hospital during the same time-period, as the probable case.
* Born within ±2 weeks from the date of birth of the case. If the list of children born within ±2 weeks is exhausted, then the range will be extended to ±4 weeks. In case a suitable control is not found even then, the range will be extended to ±6 weeks.
* Written informed consent obtained and signed from the parent or guardian of the child.

Exclusion Criteria:

For cases:

* Child has previously participated as a case or a control in this study, either in the same hospital or in another study hospital.
* Onset of SGE >48 hours after admission to the hospital (nosocomial infections).
* Child with a condition where rotavirus vaccination would be contraindicated.

For controls:

* Child has participated in the past as a case or control in this study, either in the same hospital or in another study hospital.
* Child who has symptoms of GE/ SGE during current hospital stay/ visit to the hospital outpatient clinic or on the day of interview of his/her parent or guardian.
* Child with a condition where rotavirus vaccination would be contraindicated.

Ages: 14 Weeks to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The confirmed cases are children born after 01 October 2006, at least 14 weeks of age, hospitalized for SGE during the designated study period and whose stool samples have been tested positive for RV by polymerase chain reaction (PCR). The controls are those children hospitalised or visiting the hospital outpatient clinic for non-GE causes at the study hospitals during the same time-period as the case and will be included after matching by age.
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2008-02-23 (Actual); Primary Completion 2010-06-11 (Actual); Study Completion 2010-06-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of PCR-confirmed rotavirus (RV) severe gastroenteritis (SGE) in children fully vaccinated with Rotarix or in unvaccinated children | More than 14 days after receipt of vaccine

SECONDARY OUTCOMES:
Occurrence of PCR-confirmed RV SGE in children who received one or two doses of Rotarix or in unvaccinated children | More than 14 days after receipt of vaccine
Occurrence of PCR-confirmed RV SGE in children who received at least one dose of Rotarix or Rotateq in unvaccinated children | More than 14 days after receipt of vaccine
Occurrence of SGE due to RV among children born after 01 October 2006, at least 14 weeks of age and admitted to hospital | Average time frame: 1 year from the date of subject enrolment
Occurrence of co-infections with other organisms among children born after 1 October 2006, at least 14 weeks of age and hospitalized with PCR-confirmed RV SGE | Average time frame: 1 year from the date of subject enrolment
Occurrence of PCR-confirmed RV SGE by age and month of year, among children born after 01 October 2006, at least 14 weeks of age and admitted to the hospital | Average time frame: 1 year from the date of subject enrolment
Occurrence of RV serotypes among hospitalized PCR-confirmed RV SGE children born after 01 October 2006 and at least 14 weeks of age | Average time frame: 1 year from the date of subject enrolment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- Belgium (26):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Chimay
  - GSK Investigational Site, Deinze
  - GSK Investigational Site, Deurne
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Eeklo
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Gosselies
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Heusden
  - GSK Investigational Site, Hornu
  - GSK Investigational Site, Ieper
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Merksem
  - GSK Investigational Site, Mons
  - GSK Investigational Site, Namur
  - GSK Investigational Site, Nivelles
  - GSK Investigational Site, Ostend
  - GSK Investigational Site, Ottignies
  - GSK Investigational Site, Roeselaere
  - GSK Investigational Site, Sint-Niklaas
  - GSK Investigational Site, Sint-Truiden
  - GSK Investigational Site, Tongeren
  - GSK Investigational Site, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=4240

REFERENCES:
- [Background] Braeckman T, Van Herck K, Meyer N, Pircon JY, Soriano-Gabarro M, Heylen E, Zeller M, Azou M, Capiau H, De Koster J, Maernoudt AS, Raes M, Verdonck L, Verghote M, Vergison A, Matthijnssens J, Van Ranst M, Van Damme P; RotaBel Study Group. Effectiveness of rotavirus vaccination in prevention of hospital admissions for rotavirus gastroenteritis among young children in Belgium: case-control study. BMJ. 2012 Aug 8;345:e4752. doi: 10.1136/bmj.e4752. PMID 22875947
- [Background] Braeckman T et al. Vaccine effectiveness against Community-Acquired severe Rotavirus gastroenteritis among infants, in Belgium: A hospital-based, prospective, case control study. Abstract presented at the 11th International Symposium on Double-Stranded RNA Viruses, San Juan, Puerto Rico, 27 Nov - 01 Dec 2012.
- [Background] Matthijnssens J et al. Genotype-specific vaccine effectiveness against rotavirus gastroenteritis hospitalisation among young children in Belgium. Abstract presented at the 11th International Symposium on Double-Stranded RNA Viruses, San Juan, Puerto Rico, 27 Nov - 01 Dec 2012.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111426 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111426 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111426 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111426 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111426 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111426 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register